CLINICAL TRIAL: NCT04953962
Title: Multicenter, Randomized, Parallel Group, Phase 2 to Establish the Efficacy and Safety of Combinations of CBP501, Cisplatin, and Nivolumab for ≥3rd Line Treatment of Patients With Exocrine Pancreatic Cancer and WBC <10,000/mm3 at Screening
Brief Title: Study of CBP501/Cisplatin/Nivolumab Combinations in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CanBas Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBP21-01
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer Stage IV
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cdc25C phosphatase (211-221); Cisplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: CBP501 (25) + Cisplatin + Nivolumab (Experimental): CBP501 25mg/m2 and Cisplatin 60mg/m2 will be administered simultaneously. Nivolumab 240mg will be administered following the completion of CBP501 and cisplatin infusions.
  Interventions: Drug: CBP501 (25); Drug: Cisplatin; Drug: Nivolumab
- Arm 2: CBP501 (16) + Cisplatin + Nivolumab (Experimental): CBP501 16mg/m2 and Cisplatin 60mg/m2 will be administered simultaneously. Nivolumab 240mg will be administered following the completion of CBP501 and cisplatin infusions.
  Interventions: Drug: CBP501 (16); Drug: Cisplatin; Drug: Nivolumab
- Arm 3: CBP501 (25) + Cisplatin (Experimental): CBP501 25mg/m2 and Cisplatin 60mg/m2 will be administered simultaneously.
  Interventions: Drug: CBP501 (25); Drug: Cisplatin
- Arm 4: Cisplatin + Nivolumab (Experimental): Cisplatin 60mg/m2 will be administered as infusion and then Nivolumab 240mg will be administered.
  Interventions: Drug: Cisplatin; Drug: Nivolumab

INTERVENTIONS:
Drug: CBP501 (16) — 16 mg/m2
  Other Names: CBP501
  Arms: Arm 2: CBP501 (16) + Cisplatin + Nivolumab
Drug: CBP501 (25) — 25 mg/m2
  Other Names: CBP501
  Arms: Arm 1: CBP501 (25) + Cisplatin + Nivolumab; Arm 3: CBP501 (25) + Cisplatin
Drug: Cisplatin — 60mg/m2
  Other Names: CDDP
Drug: Nivolumab — 240 mg
  Other Names: Opdivo
  Arms: Arm 1: CBP501 (25) + Cisplatin + Nivolumab; Arm 2: CBP501 (16) + Cisplatin + Nivolumab; Arm 4: Cisplatin + Nivolumab

SUMMARY:
Multicenter, randomized, open-label, parallel group phase 2 study to assess the efficacy and tolerance of four combinations of CBP501, cisplatin, and nivolumab administered once every 21 days to patients with stage IV exocrine pancreatic cancer and WBC < 10,000/mm3 at screening.

DETAILED DESCRIPTION:
Multicenter, randomized, open-label, parallel group phase 2 study to assess the efficacy and tolerance of four combinations of CBP501, cisplatin, and nivolumab administered once every 21 days to patients with stage IV exocrine pancreatic cancer and WBC < 10,000/mm3 at screening. Patients will be randomized 1:1:1:1 to the following four treatment groups, with randomization stratified by ECOG PS (0 vs 1) and liver metastasis (present vs absent):

1. CBP501 25 mg/m2 + cisplatin 60 mg/m2 + nivolumab 240 mg
2. CBP501 16 mg/m2 + cisplatin 60 mg/m2 + nivolumab 240 mg
3. CBP501 25 mg/m2 + cisplatin 60 mg/m2
4. Cisplatin 60 mg/m2 + nivolumab 240 mg No more than 4 cycles of combination therapy may be administered but patients who remain progression-free after 4 cycles may receive up to 6 additional cycle of single-agent nivolumab.

A Fleming two-stage design will be used. For each study arm, the null hypothesis that the true percentage of patients progression-free at 3 months is 10% will be tested against a one-sided alternative. In the first stage, 9 patients will be accrued to each study arm. In the first stage, if there are 1 or fewer patient progression-free at 3 months the study will be stopped for futility and if there are 4 or more patients progression-free at 3 months the study will stopped and the null hypothesis rejected. Otherwise, 14 additional patients will be accrued to the study arm for a total of 23. The null hypothesis will be rejected if 6 or more of 23 patients are progression-free at 3 months. This design yields a type I error rate of 2.5% and power of 80% when the true percentage of patients progression-free at 3 months is 35%.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to initiation of any study-specific procedures and treatment;
2. Patients with pathologically confirmed stage IV exocrine pancreatic cancer who have received at least two lines of systemic therapy for metastatic disease. Up to 10 of prior lines of systemic therapy (including prior cisplatin), chemoradiotherapy, radiotherapy or investigational agents the patient has received are allowed in order to be eligible, as long as all eligibility criteria are met, with the exception that a patient must not have received more than two prior lines incorporating anti-PD-1, anti-PD-L1, or anti-CTLA-4 immune checkpoint blockade.

   Patients who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4 immune checkpoint blockade therapy must have tolerated therapy with no evidence of grade 4 toxicity or an immune-related event (any grade) that required treatment discontinuation. Patients who experienced an endocrine related dysfunction are eligible, provided they are on stable hormone replacement therapy;
3. Male or female patients aged ≥ 18 years at time of informed consent;
4. ECOG Performance Status (PS) 0-1;
5. Life expectancy > 3 months;
6. Previous anticancer treatment must be discontinued at least 3 weeks prior to the initiation of study treatment (with the exception of 6 weeks for mitomycin C; 6 weeks for anti-androgen therapy if discontinued prior to treatment initiation, and 8 weeks for bicalutamide);
7. Adequate bone marrow reserve, cardiac, liver, renal and metabolic function:

   * white blood cell count (WBC) <10,000/mm3;
   * absolute neutrophil count (ANC) ≥ 1,500/mm3;
   * platelet count ≥ 100,000/mm3;
   * hemoglobin ≥ 9 g/dL;
   * creatinine phosphokinase isozymes CPK-MB and CPK-MM ≤ upper limit of normal (ULN);
   * serum troponin T levels within normal limits;
   * bilirubin ≤ 1.5 x ULN;
   * alanine aminotransferase (ALT, SGPT) and aspartate aminotransferase (AST, SGOT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present);
   * INR ≤ 1.5 x ULN;
   * serum creatinine ≤ ULN or creatinine clearance ≥ 60 mL/min (by Cockcroft & Gault formula or alternate calculation by 24hr urine collection). Patients with serum creatinine ≤ ULN and clearance between 45 to 59 mL/min should reduce cisplatin dose by 50%;
   * serum potassium ≥ 3.0 and ≤ 5.5 mmol/L;
   * serum calcium ≥ 8.0 and ≤ 11.5 mg/dL (≥ 2.0 and ≤ 2.9 mmol/L);
   * serum magnesium ≥ 1.2 and ≤ 3.0 mg/dL (≥ 0.5 and ≤ 1.23 mmol/L);
8. Female patients of child-bearing potential must have a negative serum pregnancy test and use at least one form of contraception as approved by the investigator for 4 weeks prior to initiating study treatment and for 14 months after the last dose of study drug . For the purposes of this study, child-bearing potential is defined as "all female patients unless they are post-menopausal for at least 3 years or surgically sterile;
9. Male patients must use a form of barrier contraception approved by the investigator during the study and for 14 months after the last dose of study drug.
10. Ability to cooperate with study treatment and follow-up.

Exclusion Criteria:

1. Radiation therapy to >30% of bone marrow prior to study entry;
2. Prior chemotherapy with nitrosoureas, prior mitomycin C cumulative dose ≥ 25 mg/m2, prior bone marrow transplant, or prior intensive chemotherapy with stem cell support;
3. Presence of any serious concomitant systemic disorders incompatible with the study in the opinion of the investigator (e.g., uncontrolled congestive heart failure, active infection, etc.);
4. Any previous history of another malignancy (other than cured basal cell or squamous cell carcinoma of the skin or cured in-situ carcinoma) within 5 years of study entry;
5. Presence of any significant central nervous system (CNS) or psychiatric disorder(s) that would hamper the patient's compliance;
6. Evidence of peripheral neuropathy grade ≥ 2;
7. Treatment with any other investigational agent or participation in another clinical trial within 28 days prior to study entry;
8. Pregnant or breast-feeding patients or any patient with child-bearing potential not using adequate contraception;
9. Known HIV, HBV, or HCV infection (excluding cured HBV and/or cured HCV infection);
10. Active CNS metastases; however, patients with CNS metastases will be eligible if they have been treated and are stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be off steroids;
11. Who require chronic systemic steroid therapy or on any other form of immunosuppressive medication;
12. Has received a live-virus vaccination within 30 days of planned treatment start;
13. With known risk factors for bowel perforation, i.e., history of diverticulitis, intra-abdominal abscess, intestinal obstruction, or abdominal carcinomatosis;
14. Has an active autoimmune disease or a documented history of autoimmune disease;
15. Has a history pneumonitis or interstitial lung disease.
16. Patients who were permanently discontinued from prior immunotherapy due to immune-related adverse events.
17. Patients who are platinum and PD-1/PD-L1 inhibitor double refractory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Three-month progression free survival rate (3M PFSR) | 3 months after treatment
  Tumor assessment by RECIST v.1.1 criteria will be performed at screening, every 8 weeks starting after Cycle 1 Day 1, at the End-of-Treatment visit, and every 3 months after the End-of-Treatment visit until disease progression is observed.

SECONDARY OUTCOMES:
Safety profiles of the combinations of CBP501, cisplatin, and nivolumab administered once every 21 days | One year
  Safety will be assessed throughout the study through clinical and laboratory safety evaluations. These include physical examinations, vital sign measurements, 12-lead ECGs, laboratory safety tests (hematology, INR, serum chemistry, serum cardiac markers), and clinical adverse experience monitoring. Adverse events will be evaluated at each visit throughout the study and assigned a grade, defined by NCI-CTCAE version 5.0 criteria, and relationship to study treatment (unrelated, related).
Progression-free survival (PFS) | one year
  Tumor assessment by RECIST v.1.1 criteria will be performed at screening, every 8 weeks starting after Cycle 1 Day 1, at the End-of-Treatment visit, and every 3 months after the End-of-Treatment visit until disease progression is observed.
Confirmed and timepoint objective response rates (cORR/ORR) | one year
  Tumor assessment by RECIST v.1.1 criteria will be performed at screening, every 8 weeks starting after Cycle 1 Day 1, at the End-of-Treatment visit, and every 3 months after the End-of-Treatment visit until disease progression is observed.
Duration of responses (DoR) | one year
  Tumor assessment by RECIST v.1.1 criteria will be performed at screening, every 8 weeks starting after Cycle 1 Day 1, at the End-of-Treatment visit, and every 3 months after the End-of-Treatment visit until disease progression is observed.
disease control rate (DCR: CR + PR + SD ≥12 weeks) | one year
  Tumor assessment by RECIST v.1.1 criteria will be performed at screening, every 8 weeks starting after Cycle 1 Day 1, at the End-of-Treatment visit, and every 3 months after the End-of-Treatment visit until disease progression is observed.
Overall survival (OS) | one year
  Tumor assessment by RECIST v.1.1 criteria will be performed at screening, every 8 weeks starting after Cycle 1 Day 1, at the End-of-Treatment visit, and every 3 months after the End-of-Treatment visit until disease progression is observed.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Arizona Oncology Associates, PC-HOPE, Tucson, Arizona
  - Ochsner Clinic Foundation, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - University of Michigan hospital, Ann Arbor, Michigan
  - Minnesota oncology Hematology, P.A., Minneapolis, Minnesota
  - James D Sanchez, Henderson, Nevada
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-McAllen South Second Street, McAllen, Texas
  - Texas Oncology- McKinney, McKinney, Texas
  - Texas Oncology-San Antonio Northeast, San Antonio, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - Texas Oncology-Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, PC, Arrington, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mine N, Yamamoto S, Kufe DW, Von Hoff DD, Kawabe T. Activation of Nrf2 pathways correlates with resistance of NSCLC cell lines to CBP501 in vitro. Mol Cancer Ther. 2014 Sep;13(9):2215-25. doi: 10.1158/1535-7163.MCT-13-0808. Epub 2014 Jul 22. PMID 25053821
- [Background] Krug LM, Wozniak AJ, Kindler HL, Feld R, Koczywas M, Morero JL, Rodriguez CP, Ross HJ, Bauman JE, Orlov SV, Ruckdeschel JC, Mita AC, Fein L, He X, Hall R, Kawabe T, Sharma S. Randomized phase II trial of pemetrexed/cisplatin with or without CBP501 in patients with advanced malignant pleural mesothelioma. Lung Cancer. 2014 Sep;85(3):429-34. doi: 10.1016/j.lungcan.2014.06.008. Epub 2014 Jul 5. PMID 25047675
- [Background] Matsumoto Y, Shindo Y, Takakusagi Y, Takakusagi K, Tsukuda S, Kusayanagi T, Sato H, Kawabe T, Sugawara F, Sakaguchi K. Screening of a library of T7 phage-displayed peptides identifies alphaC helix in 14-3-3 protein as a CBP501-binding site. Bioorg Med Chem. 2011 Dec 1;19(23):7049-56. doi: 10.1016/j.bmc.2011.10.004. Epub 2011 Oct 7. PMID 22032894
- [Background] Mine N, Yamamoto S, Saito N, Yamazaki S, Suda C, Ishigaki M, Kufe DW, Von Hoff DD, Kawabe T. CBP501-calmodulin binding contributes to sensitizing tumor cells to cisplatin and bleomycin. Mol Cancer Ther. 2011 Oct;10(10):1929-38. doi: 10.1158/1535-7163.MCT-10-1139. Epub 2011 Aug 10. PMID 21831962
- [Background] Shapiro GI, Tibes R, Gordon MS, Wong BY, Eder JP, Borad MJ, Mendelson DS, Vogelzang NJ, Bastos BR, Weiss GJ, Fernandez C, Sutherland W, Sato H, Pierceall WE, Weaver D, Slough S, Wasserman E, Kufe DW, Von Hoff D, Kawabe T, Sharma S. Phase I studies of CBP501, a G2 checkpoint abrogator, as monotherapy and in combination with cisplatin in patients with advanced solid tumors. Clin Cancer Res. 2011 May 15;17(10):3431-42. doi: 10.1158/1078-0432.CCR-10-2345. Epub 2011 Jan 10. PMID 21220472
- [Background] Sha SK, Sato T, Kobayashi H, Ishigaki M, Yamamoto S, Sato H, Takada A, Nakajyo S, Mochizuki Y, Friedman JM, Cheng FC, Okura T, Kimura R, Kufe DW, Vonhoff DD, Kawabe T. Cell cycle phenotype-based optimization of G2-abrogating peptides yields CBP501 with a unique mechanism of action at the G2 checkpoint. Mol Cancer Ther. 2007 Jan;6(1):147-53. doi: 10.1158/1535-7163.MCT-06-0371. PMID 17237275
- [Derived] Enzler T, Nguyen A, Misleh J, Cline VJ, Johns M, Shumway N, Paulson S, Siegel R, Larson T, Messersmith W, Richards D, Chaves J, Pierce E, Zalupski M, Sahai V, Orr D, Ruste SA, Haun A, Kawabe T. A multicenter, randomized phase 2 study to establish combinations of CBP501, cisplatin and nivolumab for >/=3rd-line treatment of patients with advanced pancreatic adenocarcinoma. Eur J Cancer. 2024 Apr;201:113950. doi: 10.1016/j.ejca.2024.113950. Epub 2024 Feb 22. PMID 38422585